CLINICAL TRIAL: NCT02396043
Title: Modified BFM-95 Regimen for the Treatment of Newly Diagnosed T-lymphoblastic Lymphoma in Adults:a Prospective Phase II Study
Brief Title: Modified BFM-95 Regimen as First-Line Chemotherapy in Adults With T- Lymphoblastic Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hua Wang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LBL-308
Record Dates: First submitted 2015-03-18; First posted 2015-03-24 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Lymphoma, Lymphoblastic
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Vincristine; Cyclophosphamide; Methotrexate; Mercaptopurine; Maintenance; Injections, Spinal; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Modifed BFM-95 (Experimental): All patients received induction phase 1 and phase2, followed by the protocol M, reinduction phase 1 and phase2, and maintenance (mercaptopurine 50 mg/m2 daily and methotrexate [MTX] 20 mg/m2 weekly, both orally) for up to a total therapy duration of 24 months. Response to treatment was evaluated on day 33 and at the end of induction in Modifed BFM-95.Sufficient response was defined as at least 70% tumor regression, less than 5% BM blasts, and no CNS disease on day 33 and complete remission detected by PET / CT at the end of induction.For patients with insufficient response at day 33 or at the end of induction treatment was to be intensified according to the high-risk branch of trial ALL-BFM95, with local radiotherapy (30 Gy) and allogeneic blood stem-cell transplantation.
  Interventions: Drug: induction phase1; Drug: induction phase2; Drug: protocol M; Drug: maintenance therapy; Drug: reinduction phase1; Drug: reinduction phase2; Drug: Intrathecal (IT)

INTERVENTIONS:
Drug: induction phase1 — Vincristine: 1.5 mg/m2 (max 2 mg) iv on days1, 8, 15, 22,Pirarubicin: 30 mg/m2 iv on days1, 8, 15, 22,Prednisone: 60 mg/m2 po on days 1-28.
  Pegaspargase :3750U/m2 im on days 8,22
  Other Names: Vincristine,Pirarubicin,Prednisone,Pegaspargase
Drug: induction phase2 — Cyclophosphamide: 1000 mg/m2 iv on days 35, 59,Cytarabine: 75 mg/m2 iv on days 35-38, 42-45, 49-52, 56-59,Mercaptopurine: 60 mg/m2 po on days 35-59
  Other Names: Cyclophosphamide,Cytarabine,Mercaptopurine
Drug: protocol M — Methotrexate: 5 g/m2 d 8, 22, 36, 50;Mercaptopurine:25 mg/m2 1-56
  Other Names: Methotrexate,Mercaptopurine
Drug: maintenance therapy — 6-mercaptopurine , 50 mg/m 2 daily, and Methotrexate, 20 mg/m 2 once a week.The treatment lasted 2.0 years.Note that there were four additional doses of HD-MTX(5 g/m2 ) every 3 months during the maintenance phase
  Other Names: 6-mercaptopurine,Methotrexate
Drug: reinduction phase1 — Vincristine: 1.5 mg/m2 (max 2 mg) iv on days1, 8, 15, 22,Pirarubicin: 30 mg/m2 iv on days1, 8, 15, 22,Prednisone: 60 mg/m2 po on days 1-28.
  Pegaspargase :3750U/m2 im on days 8
  Other Names: Vincristine,Pirarubicin,Prednisone,Pegaspargase
Drug: reinduction phase2 — Cyclophosphamide: 1000 mg/m2 iv on days 29,Cytarabine: 75 mg/m2 iv on days 31-34, 38-41,Mercaptopurine: 60 mg/m2 po on days 29-42
  Other Names: Cyclophosphamide,Cytarabine,Mercaptopurine
Drug: Intrathecal (IT) — methotrexate (15 mg/m 2 ), cytarabine (40 mg/m 2 ) and dexamethasone (4 mg).induction :d1, 15, 29, 45 ;Protocol M:d1, 15, 29, 43;Reinduction:d31,38
  Other Names: methotrexate ,cytarabine and dexamethasone

SUMMARY:
This study evaluates the efficacy and tolerability of treatment for T-lymphoblastic lymphoma (T-LBL) according to modified BFM-95 regimen for acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
All patients received a modified BFM regimen which was derived from the NHL-BFM-95. The differences were as follows: (1) during the course of high-dose methotrexate therapy (HD-MTX), citrovorum folinate (CF) was used for rescue at 36 h after the administration of HD-MTX;(2) Pirarubicin was used instead of daunorubicin (3) Pegaspargase was used instead of L-asparaginase for patients.All patients received induction phase 1 and phase2, followed by the protocol M, reinduction phase 1 and phase2, and maintenance (mercaptopurine 50 mg/m2 daily and methotrexate [MTX] 20 mg/m2 weekly, both orally) for up to a total therapy duration of 24 months. CNS-positive patients received two additional doses of intrathecal MTX at days 18 and 27 of induction and received CRT after reinduction therapy. The dose was 18 Gy.Patients with identifiable blasts in CSF-cytospin preparation but less than 5cells/uL in CSF were not considered CNS positive but received two additional doses of intrathecal MTX at days 18 and 27. For men with testicular involvement,orchiectomy was not performed, and irradiation (20 Gy) of testes was to be confined to biopsy-proven persistent infiltration of testis after protocol M.Response to treatment was evaluated on day 33 and at the end of induction in Modifed BFM-95.Sufficient response was defined as at least 70% tumor regression, less than 5% BM blasts, and no CNS disease on day 33 and complete remission detected by PET / CT at the end of induction.For patients with insufficient response at day 33 or at the end of induction treatment was to be intensified according to the high-risk branch of trial ALL-BFM95, with local radiotherapy (30 Gy) and allogeneic blood stem-cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosedT-LBL
* age:18-65years
* Ann Arbor stage IEto stage IVE
* at lease one measurable lesion
* receive no chemotherapy or radiotherapy before
* Adequate renal function (eg, serum creatinine≤1.5 mg/dL and creatinine clearance ≥50 mL minute), and hepatic function (e.g, total bilirubin≤ 2 times the upper limit of normal and aspartate and alanine transaminase levels ≤ 3 times the upper limit of normal)

Exclusion Criteria:

* mismatch the inclusion criteria
* systematic central nervous system involvement, previous or concomitant malignancies and any coexisting medical problems that could cause poor compliance with the study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-03; Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
progression free survival | up to end of follow-up-phase (approximately 3 years)

SECONDARY OUTCOMES:
complete remission rate | every 4 weeks,up to completion of induction treatment(approximately 2months)
overall survival | up to end of follow-up-phase (approximately 3 years)
safety, including hematological safety and non-hematological safety.All the adverse events will be classified according to Common Terminology Criteria for Adverse Events v3.0 (CTCAE) | up to end of follow-up-phase (approximately 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Hua Wang, MD., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Wang K, Chen X, Wuxiao Z, Wang Z, Sun X, Zeng Z, Li S, Xia ZJ. Long-term outcomes of modified Berlin-Frankfurt-Munster-90 regimen in adults with T-lymphoblastic lymphoma: a single-center experience. Leuk Lymphoma. 2014 Aug;55(8):1800-5. doi: 10.3109/10428194.2013.828350. Epub 2014 Mar 7. PMID 24475787